CLINICAL TRIAL: NCT03008694
Title: Phrase II Single Arm Study of Effect of FDG-PET/CT for Simulation and Radiation Treatment Planning in Oral
Brief Title: Effect of FDG-PET/CT for Simulation and Radiation Treatment Planning in Oral Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, yahua zhong, Director,oncology , Principal Investigator, Clinical Professor, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhongnanH
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Oral Cancer; Radiotherapy; Complications
Keywords: PET/CT
MeSH Terms: conditions — Mouth Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PET/CT
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — pet/ct is used as radiotherapy simulation

SUMMARY:
This study evaluates the effect of FDG-PET/CT for Simulation and Radiation Treatment Planning in oral Cancer patients. Progress-free survival (PFS) will be compared with historical control as defined in the protocol

DETAILED DESCRIPTION:
Radiotherapy improves local control and overall survival for oral cavity cancer patients after surgery. However, limited locoregional control remains a key issue in the management of oral cavity carcinomas. Appropriate target selection is a key issue in the radiotherapy of oral cavity cancer. The purpose of this study is to determine the locoregional control in PET/CT based radiotherapy treatment planning in the treatment of oral cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed oral squamous-cell carcinoma
* Age > 17 years
* Signed informed consent
* ECOG Performance status 0-2
* Must be able to start RT within 4 weeks after PET/CT simulation

Exclusion Criteria:

* stage IV disease diagnosed before acquisition of staging PET/CT
* prior radiotherapy to oral and neck
* Unable to understand study participation
* Claustrophobia
* pregnant or breast feeding mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
progress free survival | baseline to 2 years

IPD SHARING:
Plan to Share IPD: Undecided